CLINICAL TRIAL: NCT04195971
Title: Multiphasic Liver CT Scan Including Dual Arterial Phase Imaging in Patients With Liver Cirrhosis and Suspected Portal Hypertension: Evaluation of Acquisition of Appropriate Late Arterial Phase Imaging
Brief Title: Dual Arterial Phase Liver CT in Patients With Suspected Portal Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2019-2587
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: HCC; Cirrhosis, Liver
Keywords: CT
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver CT with dual arterial phase (Experimental)
  Interventions: Diagnostic Test: Liver CT

INTERVENTIONS:
Diagnostic Test: Liver CT — Liver CT with precontrast, dual arterial phase, portal venous phase, and delayed phase.

SUMMARY:
Patients with liver cirrhosis is at risk of developing HCC. To diagnose or detect HCC at CT/MRI, optimal late arterial phase (LAP) acquisition is critical to capture the tumor. For LAP acquisition, bolus-tracking is often used at CT. In patients with portal hypertension, however, bolus-tracking occasionally capture early arterial phase which may be related with slow portomesenteric flow. In this study, we obtain dual arterial phase in patients with suspected portal hypertension and determine whether this protocol (dual arterial phase) would provide higher incidence of LAP acquisition than single arterial phase acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years
* Liver cirrhosis diagnosed with characteristic imaging feature or histology
* Presence of portal hypertension sign (splenomegaly and varices)
* Scheduled for liver CT
* And signed informed consent

Exclusion Criteria:

* Relative or absolute contra-indication of contrast-enhanced CT

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of optimal late arterial phase acquisition | 1 months after study completion
  incidences of optimal late arterial phase acquisition in 1st and 2nd acquisition of arterial phase in this protocol (dual arterial phase) CT.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No